CLINICAL TRIAL: NCT04513990
Title: Evaluation of a Novel Point-of-Care Diagnostic Test for SARS-CoV-2
Brief Title: Novel Point-of-Care Diagnostic Test for SARS-CoV-2 (COVID-19)
Acronym: END CoV-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-0318; NCI-2020-03470 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0318 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-06-05; First posted 2020-08-14 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (biospecimen collection) (Experimental): Participants undergo collection of nasopharyngeal (back of the nose) samples by a medical provider and self-collection of oral, saliva, and nasal samples.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of nasopharyngeal, oral, saliva, and nasal samples
Other: Questionnaire Administration — Demographic information, sample collection type preferences; clinical outcome information

SUMMARY:
This study investigates a new diagnostic test in detecting SARS-CoV-2, the virus that causes the disease COVID-19. This may help to improve testing for COVID-19.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the clinical performance of a novel point-of-care diagnostic test for detecting severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus that causes the disease called coronavirus disease 19 (COVID-19).

SECONDARY OBJECTIVES:

I. To compare the clinical performance of provider-collected nasopharyngeal samples with self-collected nasal swab, cheek swab, and saliva sample using the novel SARS-CoV-2 diagnostic test.

II. To measure viral load and evaluate the role of viral load in COVID-19 severity.

OUTLINE:

Participants undergo collection of nasopharyngeal (back of the nose) samples by a medical provider and self-collection of oral, saliva, and nasal samples.

After completion of study, participants are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Qualifies for SARS-CoV-2 testing at MD Anderson, Lyndon B. Johnson (LBJ) hospital, or affiliated sites (may include MD Anderson and LBJ patients and employees) according to institutional criteria at time of enrollment
* Willing and able to provide informed consent
* Ability to perform protocol-required activities
* Able to speak and read English or Spanish

Exclusion Criteria:

* Patient or provider decision not to perform SARS-CoV-2 testing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of diagnostic test | Up to 1 year
  Will use the standard-of-care (real time polymerase chain reaction [RT-PCR]) coronavirus disease 19 (COVID-19) test at the MD Anderson Molecular Diagnostic Lab result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) as the true result to estimate sensitivity with 95% confidence intervals. Estimates of sensitivity and specificity of the novel point-of-care diagnostic test will be provided separately for the provider-collected nasopharyngeal samples, the self-collected nasal swab, and the self-collected cheek swab.
Specificity of diagnostic test | Up to 1 year
  Will use the standard-of-care (RT-PCR) COVID-19 test at the MD Anderson Molecular Diagnostic Lab result for SARS-CoV-2 as the true result to estimate specificity with 95% confidence intervals. Estimates of sensitivity and specificity of the novel point-of-care diagnostic test will be provided separately for the provider-collected nasopharyngeal samples, the self-collected nasal swab, and the self-collected cheek swab.
Concordance of the novel point-of-care diagnostic test | Up to 1 year
  Will be estimated with 95% confidence intervals.
Positive predictive value (PPV) of the novel point-of-care diagnostic test | Up to 1 year
  Will be estimated with 95% confidence intervals.
Negative predictive value (NPV) of the novel point-of-care diagnostic test | Up to 1 year
  Will be estimated with 95% confidence intervals.

SECONDARY OUTCOMES:
Viral load metrics | Up to 1 month
  Will use descriptive statistics to summarize viral load metrics from the standard-of-care (RT-PCR) SARS-CoV-2 test and from each of the point-of-care tests.
Disease progression | Up to 1 month
  Will use logistic regression methods to model progression to severe disease (defined as hospitalization) as a function of viral load, age, gender, smoking history, comorbidities, and symptoms for each of these tests.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Schmeler, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org